CLINICAL TRIAL: NCT05905562
Title: Effects of Core Muscle Activation Exercise Training Program on Pain, Range of Motion, and Function in Patients With Chronic Low Back Pain
Brief Title: Core Muscle Activation Exercise Training Program Effects in Patients With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0114
Record Dates: First submitted 2023-04-18; First posted 2023-06-15 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spinal mobilization and core stabilization exercises group: (Experimental): will have core muscle activation exercises along with lumber spine joint mobilization along with TENS and Ultrasound for 12 weeks and 3 sessions per week
  Interventions: Other: core stabilization exercises; Other: Spinal mobilization techniques
- Spinal mobilization techniques group (Active Comparator): will have lumber spine joint mobilization along with TENS and Ultrasound duration of 12 weeks with 3 sessions per week.
  Interventions: Other: Spinal mobilization techniques

INTERVENTIONS:
Other: core stabilization exercises — Core muscles activation exercises will be performed on patients to target the abdominals.
  Arms: Spinal mobilization and core stabilization exercises group:
Other: Spinal mobilization techniques — lumbar spine joint mobilization techniques will be performed to patient in prone lying.

SUMMARY:
The study will be a Randomized clinical trial to check the effects of a core muscle activation exercise training program on pain, range of motion, and function in patients with chronic low back pain so that we can devise a treatment protocol for patients with chronic low back pain. The study duration was 10 months, convenient sampling technique was used subject following eligibility criteria from the Orthopaedic medical center, Lahore. were randomly allocated in two groups via lottery method, a baseline assessment was done, and Group A received Mobilization and Electrotherapy Modalities including Ultrasound, TENS, and Core muscles activation exercises. Group B received Mobilization and Electrotherapy Modalities including Ultrasound and TENS for a total training program duration of 12 weeks with 3 sessions per week. Outcome measures were NPRS for assessment of pain, Modified Oswestry Disability index for functional disability, PBU for assessment and training of core stability, and baseline bubble inclinometer and were assessed and documented at 0 week, 4 weeks, 8 weeks, and 12 weeks of the treatment session

DETAILED DESCRIPTION:
Low back pain is one of the most common musculoskeletal disorders in both males and females, with a prevalence rate of 80% of the world population. However, in some cases, acute low back pain persists for more than 3 months and becomes chronic low back pain. During low back pain, significant complaints of patients other than pain are decreased mobility and functional limitations in their workplace and at home In recent years, multiple studies have explored the evidence for treating chronic low back pain; options include soft tissue mobilization, spinal manipulation therapy, spinal joint mobilization therapy, behavioral therapy, exercise therapy, transcutaneous electrical nerve stimulation, interferential currents, low-level laser therapy, and yoga. Other treatments include massage, acupuncture, and superficial heat therapy thermal heat wraps, hot water bottles, heated packs filled with grain, hot towels, and electric heating pads). Manual modalities such as physiotherapy, massage, chiropractic, occupational, and osteopathic therapies, including spinal manipulation and mobilization, are often used together and alone to treat chronic non-specific low back pain Exercises are a way to induce strength, endurance, functional mobility, and neuromuscular control in back muscles. A variety of Exercises like Motor control stabilization exercises, back stabilization exercises, core muscle activation exercises, and endurance exercises are used to reduce the effect of low back pain. These particular exercises are for lumber and core Stabilization and strengthening but there is very limited research on the superiority of each exercise over the other.

Earlier work suggested that there is little or no evidence that spinal manipulative therapy was superior to other standard treatments for chronic low back pain. however, recent systematic reviews suggest that spinal manipulation and mobilization are "viable" options for pain treatment

ELIGIBILITY:
Inclusion Criteria:

* • Both Gender

  * Age range from 20-50 years.
  * Chronicity of low back pain for at least 3 months.

Exclusion Criteria:

* Patients with any signs of spinal cord involvement
* Pregnant female patients
* History of spinal trauma or spinal or abdominal surgery
* History of systemic disease (e.g., systemic scleroderma or muscular dystrophy), spinal deformity (e.g., scoliosis and kyphosis), or abdominal wall hernia
* History of participation in core stability exercise or any physical therapy treatment in the past 6 months
* Any bony or soft tissue systemic disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Bubble base inclinometer for Range of Motion | up to 12 weeks
  It will be used to measure lumbar Range of motion. It will be placed near the joint to be measured; turn the dial until the scale reads zero; take the joint through its range and range of motion will be recorded (in degrees) directly from the dial.
Pressure biofeedback unit for Muscle strength | up to 12 weeks
  Pressure Biofeedback Unit will be use to assess core stability muscle strength contraction. pressure biofeedback unit will be placed under the lumbar spine at the height of L3 and inflate the cuff to 40mmHg.The patient is then instructed to perform core contraction and increase the pressure in steps of 2-4mmHg. So from 40 to 42or44mmHg and so on. The contraction should be held whilst being able to keep breathing calmly. Ideally, the patient is able to hold this contraction for 15 seconds. Time will be noted.
Numeric Pain Rating Scale | up to 12 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes
Modified Oswestry Disability Index | up to 12 weeks
  The Oswestry Disability Index (also known as the Oswestry Low Back Pain Disability Questionnaire) is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. It has 10 different sections. For each section the total possible score is 5. If all 10 sections are completed the score is calculated and interpreted in percentage measures.

CONTACTS AND LOCATIONS:
Overall Officials: Sana Gohar, MS*, Principal Investigator — Riphah International University
Locations (1):
- Orthopedics Medical Complex Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Coulter ID, Crawford C, Hurwitz EL, Vernon H, Khorsan R, Suttorp Booth M, Herman PM. Manipulation and mobilization for treating chronic low back pain: a systematic review and meta-analysis. Spine J. 2018 May;18(5):866-879. doi: 10.1016/j.spinee.2018.01.013. Epub 2018 Jan 31. PMID 29371112
- [Background] Waseem M, Karimi H, Gilani SA, Hassan D. Treatment of disability associated with chronic non-specific low back pain using core stabilization exercises in Pakistani population. J Back Musculoskelet Rehabil. 2019;32(1):149-154. doi: 10.3233/BMR-171114. PMID 30248035
- [Background] Areeudomwong P, Buttagat V. Comparison of Core Stabilisation Exercise and Proprioceptive Neuromuscular Facilitation Training on Pain-related and Neuromuscular Response Outcomes for Chronic Low Back Pain: A Randomised Controlled Trial. Malays J Med Sci. 2019 Nov;26(6):77-89. doi: 10.21315/mjms2019.26.6.8. Epub 2019 Dec 30. PMID 31908589
- [Background] Ozsoy G, Ilcin N, Ozsoy I, Gurpinar B, Buyukturan O, Buyukturan B, Kararti C, Sas S. The Effects Of Myofascial Release Technique Combined With Core Stabilization Exercise In Elderly With Non-Specific Low Back Pain: A Randomized Controlled, Single-Blind Study. Clin Interv Aging. 2019 Oct 9;14:1729-1740. doi: 10.2147/CIA.S223905. eCollection 2019. PMID 31631992
- [Background] Mueller J, Niederer D. Dose-response-relationship of stabilisation exercises in patients with chronic non-specific low back pain: a systematic review with meta-regression. Sci Rep. 2020 Oct 9;10(1):16921. doi: 10.1038/s41598-020-73954-9. PMID 33037280
- [Background] Frizziero A, Pellizzon G, Vittadini F, Bigliardi D, Costantino C. Efficacy of Core Stability in Non-Specific Chronic Low Back Pain. J Funct Morphol Kinesiol. 2021 Apr 22;6(2):37. doi: 10.3390/jfmk6020037. PMID 33922389
- [Background] Hlaing SS, Puntumetakul R, Khine EE, Boucaut R. Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 30;22(1):998. doi: 10.1186/s12891-021-04858-6. PMID 34847915
- [Background] Kumar T, Kumar S, Nezamuddin M, Sharma VP. Efficacy of core muscle strengthening exercise in chronic low back pain patients. J Back Musculoskelet Rehabil. 2015;28(4):699-707. doi: 10.3233/BMR-140572. PMID 25467999
- [Background] Sanchez Romero EA, Fernandez Carnero J, Villafane JH, Calvo-Lobo C, Ochoa Saez V, Burgos Caballero V, Laguarta Val S, Pedersini P, Pecos Martin D. Prevalence of Myofascial Trigger Points in Patients with Mild to Moderate Painful Knee Osteoarthritis: A Secondary Analysis. J Clin Med. 2020 Aug 7;9(8):2561. doi: 10.3390/jcm9082561. PMID 32784592